CLINICAL TRIAL: NCT05931393
Title: Phase 2, Open-label, Single Cohort, Multicenter Trial for Sequential Treatment of High Dose Cabozantinib on/After Progression on Cabozantinib Monotherapy in Advanced Renal Cell Carcinoma (Seq-Cabo)
Brief Title: Sequential Treatment of Cabozantinib for Advanced Renal Cell Carcinoma (RCC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Tian Zhang, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0439
Record Dates: First submitted 2023-06-22; First posted 2023-07-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: RCC; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cabozantinib Dose Escalation (Experimental): cabozantinib 80mg PO daily
  Interventions: Drug: Cabozantinib 80 MG

INTERVENTIONS:
Drug: Cabozantinib 80 MG — cabozantinib 80mg daily

SUMMARY:
The goal of this clinical trial is to learn about the effects of a higher dose of ncabozantinib in patients with advanced renal cell carcinoma who have progressed on or after receiving cabozantinib treatment.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single cohort, phase II study to assess the efficacy of cabozantinib dose escalation at the time of progression on/after cabozantinib monotherapy. The study will enroll subjects with advanced RCC (defined as locally advanced, unresectable or metastatic) who have disease progression on/after cabozantinib monotherapy in any line of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced RCC (defined as locally advanced unresectable or metastatic) of any histology who progressed on/after cabozantinib monotherapy in any line of treatment. Patient must have cabozantinib sensitive disease (prior treatment with cabozantinib ≥ 6 months)
2. Ability to tolerate prior cabozantinib at 60mg PO daily with manageable toxicity profile at the respective doses, at investigator discretion
3. Prior PD-1 inhibitor/PD-L1 inhibitor allowed
4. Evidence of measurable disease per RECIST 1.1
5. For up to 5 patients opting into on-treatment biopsy, one of the following must be met:

   1. Archival tissue confirmed to be available and obtained within 30 days of informed consent as well as willingness to undergo an on-treatment biopsy at 12 weeks (+/- 7 days).

      OR
   2. Willingness to undergo a baseline biopsy prior to Cycle 1 Day1, as well as an on-treatment biopsy at 12 weeks (+/- 7 days).
6. Age ≥ 18 at time of consent
7. ECOG performance status ≤ 2
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document
9. No washout period is needed for cabozantinib, minimum of 4 weeks or 4 half-lives washout, whichever is shorter, for other standard or experimental anti-cancer therapies.
10. Recovery to baseline or ≤ Grade 1 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy
11. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

    1. Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor (G-CSF) support
    2. White blood cell (WBC) count ≥ 2500/µL
    3. Platelets ≥ 100,000/µL without transfusion
    4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L) (transfusion acceptable per investigator discretion)
    5. Alanine transaminase (ALT), AST and alkaline phosphatase (ALP) ≤ 3 x ULN. ALP ≤ 5x ULN with documented bone metastases
    6. Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3x ULN)
    7. Serum albumin ≥ 2.8 g/dl
    8. Prothrombin (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test < 1.3x the laboratory ULN
    9. Serum creatinine ≤ 1.5x ULN or calculated creatinine clearance ≥ 40mL/min (≥ 0.675mL/sec) using the Cockcroft-Gault equation:

       * Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)
       * Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
    10. Urine protein/creatinine ratio (UPCR) ≤1 mg/mg (≤113.2 mg/mmol), or 24h urine protein ≤1 g
12. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of cabozantinib

Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

1. Female subjects are considered to be of childbearing potential unless one of the following criteria is met:

   * documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or
   * documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes.
2. In addition, females < 55 years-of-age must have a serum follicle stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause.

Exclusion Criteria:

1. Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible
2. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for 1) at least 2 weeks after radiotherapy or 2) at least 4 weeks after major surgery (e.g., removal or biopsy of brain metastasis) prior to first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment for the brain metastasis at the time of first dose of study treatment
3. Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following: 1) prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH). 2) Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
4. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   1. Cardiovascular disorders: 1) congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias; 2) uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 1 week of treatment; 3) stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis [DVT], pulmonary embolism [PE]) within 6 months before first dose of study treatment. Note: subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #3.2.4) for at least 1 week before first dose of study treatment
   2. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation, including 1) the subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction; 2) abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment
5. Clinically significant hematuria, hematemesis, hemoptysis, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 6 weeks before first dose of study treatment. (Clinically significant hematuria defined by needing transfusion; clinically significant hematemesis or hemoptysis defined by needing hospital admission)
6. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation. Cavitary pulmonary lesions are allowed if not symptomatic.
7. Lesions invading or encasing any major blood vessels
8. Other clinically significant disorders that would preclude safe study participation

   1. Serious non-healing wound/ulcer/bone fracture
   2. Moderate to severe hepatic impairment (Child-Pugh B or C).
   3. Acute COVID-19 infection - clinical recovery from COVID-19 infection at least 14 days prior to enrollment allowed.
9. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
10. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 14 days before first dose of study treatment. Furthermore, subjects with a history of additional risk factors for torsades de pointes (e.g., long QT syndrome) are also excluded. Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
11. Pregnant or lactating females
12. Inability to swallow tablets
13. Previously identified allergy or hypersensitivity to components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded
14. Another malignancy within 2 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, Gleason 6 prostate cancer, or carcinoma in situ of cervix or breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival of cabozantinib | From time of enrollment/treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason up to 24 months
  Progression free survival (PFS) will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST v 1.1)

SECONDARY OUTCOMES:
Objective Response Rate of cabozantinib | Follow up until disease progression, up to 24 months.
  To determine the Objective Response Rate (including stable disease/partial response/complete response) of of cabozantinib or cabozantinib-nivolumab combination assessed by RECIST (version 1.1)
Disease Control Rate of of cabozantinib | Follow up until disease progression, up to 24 months.
  To determine the disease control rate (including stable disease/partial response/complete response) of of cabozantinib or cabozantinib-nivolumab combination assessed by RECIST (version 1.1)
Duration of response of of cabozantinib | Follow up until disease progression, up to 24 months.
  To determine the duration of response of of cabozantinib or cabozantinib-nivolumab combination compared to historical controls assessed by RECIST (version 1.1)
Overall survival of of cabozantinib | Follow up until death or withdrawal, up to 36 months.
  To determine the overall survival rate of response of of cabozantinib or cabozantinib-nivolumab combination compared to historical controls assessed by RECIST (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Tian Zhang, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States